CLINICAL TRIAL: NCT02950779
Title: An Investigation Into Handgrip Strength as a Dietetic Assessment Tool to Detect Changes in the Nutritional and Health Status of Adults With Inflammatory Bowel Disease: A Longitudinal Observational Pilot Study
Brief Title: Assessment of Handgrip Strength in Adults With Inflammatory Bowel Disease
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: University of Southampton (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other)
Responsible Party: Sponsor
Other Study IDs: RHM MED1346
Record Dates: First submitted 2016-10-28; First posted 2016-11-01 (Estimated); Last update posted 2016-11-01 (Estimated); Status verified 2016-10

CONDITIONS: Inflammatory Bowel Disease; Nutrition
MeSH Terms: conditions — Inflammatory Bowel Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: Handgrip Strength Measurement

SUMMARY:
Inflammatory bowel disease (IBD) is a chronic disease, which causes inflammation of the gut. People with this disease are often poorly nourished. Problems caused by poor nutrition such as poor wound healing can be reduced if it is recognised and treated early.

When people with IBD attend outpatients clinic with their IBD specialist they are weighed and their BMI calculated to indicate if they are poorly nourished. Weight and BMI may not always provide a good assessment of how well nourished a person is because it does not describe the amount of muscle in the body in proportion to fat. A person with a low or decreasing amount of muscle but a normal or high BMI is at risk of nutritional problems. Measuring the amount of muscle someone with IBD has in routine practice poses a challenge to clinicians due to time constraints. One-way of measuring the amount of muscle a person has is to measure their muscle strength. This can be measured by recording the strength of a person's handgrip. Handgrip strength can be measured using a hand-held device called a dynamometer.

This study aims to test whether it is possible to measure the handgrip strength of people with IBD attending outpatient's clinic. It also aims to test how the measure obtained compares with other methods of assessing whether someone is malnourished and their health. People with a diagnosis of IBD who are aged 18 or older and who are scheduled to attend IBD outpatients clinic in one hospital will be asked to take part in the study. Their handgrip strength will be measured each time they attend clinic over a nine-month period in addition to other information about their health and nutritional state. This study forms part of a Masters in Research being undertaken with The University of Southampton.

ELIGIBILITY:
Inclusion Criteria:

1. Adult participants with a confirmed diagnosis of IBD (≥18 years of age)
2. People deemed to have capacity to consent
3. People able to understand and read English
4. People attending a gastroenterology outpatient clinic appointment

Exclusion Criteria:

1. People physically unable to complete the study procedures
2. Any person who is currently participating in another research trial in which the principle investigator is not satisfied to sign a 12-week exemption form.
3. People involved in an interventional study.
4. People who are currently an inpatient

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult participants with Inflammatory Bowel Disease attending the Gastroenterology Clinic
Sampling Method: Probability Sample
Enrollment: 25 (Estimated)
Dates: Start 2016-10; Primary Completion 2017-08 (Estimated); Study Completion 2017-10 (Estimated)

PRIMARY OUTCOMES:
Handgrip strength measurement | 12 months

SECONDARY OUTCOMES:
IBD Disease activity | 12 months
Quality of life Assessment | 12 Months
Physical Activity Assessment | 12 months
Malnutrition Screening score | 12 months
Micronutrient values | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Fraser Cummings, Dr, Study Chair — University Hospital Southampton NHS Foundation Trust

IPD SHARING:
Plan to Share IPD: No